CLINICAL TRIAL: NCT00045045
Title: A Study Of 18 FDG PET In The Prediction Of Relapse In Patients With A Clinical Stage I Non-Seminomatous Germ Cell Tumor
Brief Title: Positron Emission Tomography in Detecting Testicle Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: CDR0000256314; MRC-TE22; EU-20115
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-09

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage I malignant testicular germ cell tumor; testicular choriocarcinoma; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Carcinoma, Embryonal; Seminoma; Teratoma; Endodermal Sinus Tumor; Teratoma, Testicular | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Imaging procedures such as positron emission tomography may improve the ability to detect the extent of cancer and allow doctors to plan more effective treatment for patients who have testicle cancer.

PURPOSE: Diagnostic trial to study the effectiveness of positron emission tomography using fludeoxyglucose F 18 in predicting relapse in patients who have stage I germ cell tumor of the testicle.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the ability of fludeoxyglucose F 18 positron emission tomography to predict relapse requiring adjuvant chemotherapy in patients with high-risk stage I non-seminomatous or mixed seminoma/non-seminomatous germ cell tumor of the testis who are on current management protocols.

OUTLINE: This is a multicenter study.

Patients receive fludeoxyglucose F 18 (FDG) IV followed 1 hour later by positron emission tomography (PET) imaging. Patients with metastatic disease identified by FDG PET imaging may receive adjuvant chemotherapy according to the standard clinical practice at each participating center. Patients with no metastatic disease identified by FDG PET imaging are considered for entry into the MRC-TE08 trial (randomized trial of 2 CT scan frequencies in the surveillance of stage I teratoma) or are followed according to the standard surveillance schedule.

Patients with metastatic disease are followed every 6 months. Patients with no metastatic disease are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, and then every 4-6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 135 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-seminomatous or mixed seminoma/non-seminomatous germ cell tumor of the testis with evidence of vascular (lymphatic or venous) invasion in primary specimen
* Clinical stage I on the basis of clinical examination, chest x-ray, and CT scan of the chest, abdomen, and pelvis
* Negative post-orchidectomy tumor markers (alpha-fetoprotein and beta human chorionic gonadotropin)
* High-risk disease

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No evidence of active inflammatory or infective diseases
* No other disease or prior malignancy that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No more than 8 weeks since prior orchidectomy

Other

* No prior positron emission tomography scans

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-05; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Huddart, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - Royal Devon and Exeter Hospital, Exeter, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Guy's and St. Thomas' Hospitals NHS Foundation Trust, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Result] Huddart RA, O'Doherty MJ, Padhani A, Rustin GJ, Mead GM, Joffe JK, Vasey P, Harland SJ, Logue J, Daugaard G, Hain SF, Kirk SJ, MacKewn JE, Stenning SP; NCRI Testis Tumour Clinical Study Group. 18fluorodeoxyglucose positron emission tomography in the prediction of relapse in patients with high-risk, clinical stage I nonseminomatous germ cell tumors: preliminary report of MRC Trial TE22--the NCRI Testis Tumour Clinical Study Group. J Clin Oncol. 2007 Jul 20;25(21):3090-5. doi: 10.1200/JCO.2006.09.3831. PMID 17634488